CLINICAL TRIAL: NCT03920280
Title: Clinical Evaluation of a Daily Wear Frequent Replacement Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-C009
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Refractive Errors
Keywords: Contact Lens; Daily Wear; Vision Correction
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID015385 (Experimental): LID015385 contact lenses worn in both eyes during waking hours only for at least 8 hours per day and 5 days per week over a 3-month exposure period. Lenses will be removed nightly for cleaning with CLEAR CARE.
  Interventions: Device: LID015385 contact lenses; Device: CLEAR CARE
- Biofinity (Active Comparator): Comfilcon A contact lenses worn in both eyes during waking hours only for at least 8 hours per day and 5 days per week over a 3-month exposure period. Lenses will be removed nightly for cleaning with CLEAR CARE.
  Interventions: Device: Comfilcon A soft contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: LID015385 contact lenses — Investigational silicone hydrogel contact lenses
  Arms: LID015385
Device: Comfilcon A soft contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Biofinity
  Arms: Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based cleaning and disinfecting system

SUMMARY:
The purpose of this clinical study is to demonstrate the safety and performance of an investigational soft contact lens compared to a commercially available soft contact lens when worn in a daily wear modality.

DETAILED DESCRIPTION:
Subjects will be randomized to wear either the investigational contact lenses or the commercially available contact lenses in both eyes. Subjects will be expected to attend 6 scheduled study visits. Individual participation in the study will be approximately 3 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Manifest cylinder ≤ 0.75 diopter (D) in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Monovision contact lens wearers.
* Habitually wearing Biofinity® lenses.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6355, Orlando, Florida
  - Alcon Investigator 6291, Pensacola, Florida
  - Alcon Investigator 3950, Bloomington, Illinois
  - Alcon Investigator 6567, Pittsburg, Kansas
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 6401, Warwick, Rhode Island
  - Alcon Investigator 6353, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 investigative sites located in the United States.
Pre-assignment Details: Of the 120 subjects enrolled, 1 was exited from the study prior to randomization as a screen failure. This reporting group includes all enrolled and dispensed subjects (119).
Units Other Than Participants: eyes
Groups:
- Biofinity: Comfilcon A contact lenses worn in both eyes during waking hours only for at least 8 hours per day and 5 days per week over a 3-month exposure period. Lenses were removed nightly for cleaning with CLEAR CARE.
- LID015385: LID015385 contact lenses worn in both eyes during waking hours only for at least 8 hours per day and 5 days per week over a 3-month exposure period. Lenses were removed nightly for cleaning with CLEAR CARE.
Period: Overall Study
Arm/Group | Biofinity | LID015385
Started | 41; 82 eyes | 78; 156 eyes
Completed | 38; 76 eyes | 72; 144 eyes
Not Completed | 3; 6 eyes | 6; 12 eyes
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Corneal cylinder greater than 1.00 diopter | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled and dispensed subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofinity | LID015385 | Total
Number analyzed (Participants) | 41 | 78 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.7) | 32.9 (7.7) | 32.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 63 | 91
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 40 | 74 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 39 | 67 | 106
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 41 | 78 | 119

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses - Completed Eyes
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 1 Dispense; Week 1 Follow-up; Week 2 Follow-up; Month 1 Follow-up; Month 2 Follow-up; Month 3 Follow-up/Exit (at least 4 hours after lens insertion at each follow-up assessment visit)
Population: This analysis population includes all enrolled and dispensed subjects/eyes that completed the study.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 38 | 72
Number analyzed (eyes) | 76 | 144
logMAR
  Day 1 Dispense | -0.06 (0.06) | -0.06 (0.06)
  Week 1 Follow-up | -0.06 (0.06) | -0.05 (0.06)
  Week 2 Follow-up | -0.06 (0.06) | -0.06 (0.06)
  Month 1 Follow-up | -0.06 (0.06) | -0.05 (0.06)
  Month 2 Follow-up | -0.05 (0.06) | -0.04 (0.06)
  Month 3 Follow-up/Exit | -0.05 (0.06) | -0.05 (0.06)

2. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses - Discontinued Eyes
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen and converted to the logarithm minimum angle of resolution (logMAR) scale. A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 1 Dispense; Week 1 Follow-up; Week 2 Follow-up; Month 1 Follow-up; Month 2 Follow-up (at least 4 hours after lens insertion at each follow-up assessment visit)
Population: This analysis population includes all enrolled and dispensed subjects/eyes that discontinued the study early.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 3 | 6
Number analyzed (eyes) | 6 | 12
logMAR
  Day 1 Dispense | -0.04 (0.06) | -0.06 (0.07)
  Week 1 Follow-up: number analyzed (Participants) | 3 | 5
  Week 1 Follow-up: number analyzed (eyes) | 6 | 10
  Week 1 Follow-up | -0.02 (0.05) | -0.06 (0.07)
  Week 2 Follow-up: number analyzed (Participants) | 3 | 5
  Week 2 Follow-up: number analyzed (eyes) | 6 | 10
  Week 2 Follow-up | -0.04 (0.06) | -0.05 (0.06)
  Month 1 Follow-up: number analyzed (Participants) | 2 | 1
  Month 1 Follow-up: number analyzed (eyes) | 4 | 2
  Month 1 Follow-up | 0.00 (0.00) | -0.12 (0.00)
  Month 2 Follow-up: number analyzed (Participants) | 0 | 1
  Month 2 Follow-up: number analyzed (eyes) | 0 | 2
  Month 2 Follow-up |  | -0.12 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 3 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all enrolled and dispensed subjects.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- Biofinity - Ocular; Biofinity - Nonocular/Systemic: Events reported in this group occurred while exposed to the comfilcon A contact lenses
- LID015385 - Ocular; LID015385 - Nonocular/Systemic: Events reported in this group occurred while exposed to the LID015385 contact lenses
Arm/Group | Pretreatment | Biofinity - Ocular | Biofinity - Nonocular/Systemic | LID015385 - Ocular | LID015385 - Nonocular/Systemic
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/82 | 0/41 | 0/156 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/119 | 1/82 | 0/41 | 0/156 | 0/78
Other Adverse Events (participants affected / at risk) | 0/119 | 0/82 | 0/41 | 0/156 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=119) | Biofinity - Ocular (N=82) | Biofinity - Nonocular/Systemic (N=41) | LID015385 - Ocular (N=156) | LID015385 - Nonocular/Systemic (N=78)
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03920280/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03920280/SAP_001.pdf